CLINICAL TRIAL: NCT03160573
Title: Efficacy of ClōSYS Oral Rinse Products in Human Subjects in Controlling Oral Malodor
Brief Title: Controlling Oral Malodor by ClōSYS Oral Rinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowpar Pharmaceuticals, Inc. (Industry)
Collaborators: University Health Resources Group, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UHRG-RPR-Malodor-ADA-2016
Record Dates: First submitted 2017-05-10; First posted 2017-05-19 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Oral Malodor
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Test-Unflavored Rinse then Placebo Unflavored Rinse (Active Comparator): Participants will receive CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution for 3 weeks,. After a washout period of 2 weeks, they will then receive Placebo unflavored rinse containing containing NO 0.1% stabilized chlorine dioxide for 3 weeks.
  Interventions: Drug: ClōSYS® Unflavored Rinse
- Test-Flavored Rinse then Placebo Flavored Rinse (Active Comparator): Participants will receive CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution for 3 weeks. After a washout period of 2 weeks, they will then receive Placebo flavored rinse containing NO 0.1% stabilized chlorine dioxide for 3 weeks.
  Interventions: Drug: ClōSYS® Flavored Rinse
- Flavored Oral Rinse-Placebo then Test-Flavored Rinse (Placebo Comparator): Participants will receive CloSYS mint flavored rinse containing NO 0.1% stabilized chlorine dioxide for 3 weeks. After a washout period of 2 weeks, they will then receive CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution for 3 weeks.
  Interventions: Other: Placebo-Flavored Oral Rinse
- Unflavored Oral Rinse-Placebo then Test-Unflavored Rinse (Placebo Comparator): Participants will receive CloSYS unflavored rinse containing NO 0.1% stabilized chlorine dioxide for 3 weeks. After a washout period of 2 weeks, they will then receive unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution for 3 weeks.
  Interventions: Other: Placebo-Unflavored Oral Rinse

INTERVENTIONS:
Drug: ClōSYS® Unflavored Rinse
  Other Names: Mouth rinse
  Arms: Test-Unflavored Rinse then Placebo Unflavored Rinse
Drug: ClōSYS® Flavored Rinse
  Other Names: Mouth rinse
  Arms: Test-Flavored Rinse then Placebo Flavored Rinse
Other: Placebo-Flavored Oral Rinse — Flavor-matched placebo rinse
  Arms: Flavored Oral Rinse-Placebo then Test-Flavored Rinse
Other: Placebo-Unflavored Oral Rinse — Unflavored-matched placebo rinse
  Arms: Unflavored Oral Rinse-Placebo then Test-Unflavored Rinse

SUMMARY:
The purpose of this Study is to assess the efficacy of two ClōSYS Oral Rinse products in human subjects in controlling oral malodor in partial fulfillment of the requirements for recognition by the American Dental Association's (ADA) requirement for obtaining ADA Seal for malodor.

DETAILED DESCRIPTION:
Study Design:

The products used in this study are: ClōSYS Alcohol-Free Oral Rinse (referred here as ClōSYS Unflavored Oral Rinse) and ClōSYS justRIGHT MILD MINT Oral Rinse (referred here as ClōSYS Flavored Oral Rinse). This is an in-vivo, eight-week, a single-center, randomized, double-blind (subject/investigator), 2-waycross-overdesign clinical study. There will be two independent groups. Each subject of each group will be crossed over to the other group within a same group after the washout period. Each group will have their own control group. In the first phase, 25 subjects (50%) of each group will randomly be assigned to the active group; the other 25 subjects will be assigned to the control group. In the second phase, the participants will be crossed over of group assignment. The Study will enroll 100 subjects, aged 21 to 65 years, with a slight to strong intrinsic oral malodor, as determined by a panel of trained odor judges calibrated and standardized using a range of standard odorants sufficient to reflect the different patterns of nose receptors.

Study Plan:

Subjects will receive verbal and written oral hygiene instructions, and either one bottle (16 oz. each) of ClōSYS Unflavored Oral Rinse, ClōSYS Flavored Oral Rinse- or Placebo Oral Rinse each week. Subjects will also receive measuring cups for dispensing the rinse and a diary log for recording usage (the Oral Hygiene Kit) for use during the treatment. After a 2-week wash out period, each subject will receive another bottle of oral rinse according to their group assignment. The rinse bottles will be weighed prior to dispensing the product. A product log will be maintained and the weights of the bottles will be documented at each visit.

Subjects will be instructed to rinse twice a day, each in the morning and in the evening, with 15 mL mouth rinse for 30 seconds. They will note in their patient's log the date and time of rinsing.

Subjects will be instructed to continue with their normal oral hygiene practices, including tooth brushing and flossing but omitting any use of oral rinses or mouthwashes except for the Study materials. The subjects also will be instructed not to use other non-study related products such as breath mints, lozenge, gums, etc. as well as refraining from elective dental procedures during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read, signed, and received a copy of the Informed Consent prior to Study initiation.
2. Subject is able to follow verbal and/or written instructions, perform oral hygiene procedures and return to the test facility for specified Study examinations.
3. Subject is between the ages of 21 and 65 years of age, male or female.
4. Subject has normal oral interior cheek wall tissues.
5. Subject is in good general health as determined by medical history and clinical judgment that no severe or debilitating disease exists that would impede participation in the Study.
6. Subject must have an average organoleptic intensity rating of at least 2.6 but maximum 4.5 on an intensity scale of 0-5.

Exclusion Criteria:

1. Pregnant or nursing per subject report.
2. Diagnosis of Xerostomia, including medication induced Xerostomia.
3. Any oral or extraoral piercing that interferes with the ability to perform study procedures and/or clinical assessments in the mouth.
4. Fixed or removable oral appliance, such as orthodontic brackets or retainer, partial or complete dentures.
5. Have advanced periodontal disease or excessive gingival recession, per Investigator/Examiner discretion.
6. A known allergy or sensitivity to products planned for use in this study.
7. Unwillingness to abstain from all other oral hygiene products other than those prescribed for the duration of the study.
8. Heavy deposits of calculus, either supragingival and/or subgingival, per Investigator/Examiner discretion.
9. Have a history of severe transmittable infectious disease (hepatitis, HIV, tuberculosis).
10. Have a medical or dental condition that would be unduly affected by participation in this study, per Investigator discretion.
11. Any other condition that Principal Investigator would consider interfering with the study.
12. Smokers.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nachnani, Ph.D., Principal Investigator — University Health Resources Group, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: United Health Resources Group (UHRG) was responsible for recruitment using advertising and volunteers from their website. All patients were recruited at a single UHRG site (7721 S. Painter Ave, Whittier, CA 90602)
Pre-assignment Details: No significant events prior to assignment to an arm.
Groups:
- Test-Unflavored Rinse Then Placebo-Unflavored Rinse: CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Unflavored Rinse: Subjects in Test group will receive ClōSYS® Unflavored Rinse then Placebo-Unflavored rinse
- Test-Flavored Rinse Then Placebo-Flavored Rinse: CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Flavored Rinse: Subjects in Test group will receive ClōSYS® Flavored Rinse then Placebo Flavored Rinse
- Flavored Oral Rinse-Placebo Then Test-Flavored Rinse: CloSYS mint flavored rinse containing NO 0.1% stabilized chlorine dioxide
  Flavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Flavored Rinse then CloSYS mint flavored rinse containing 0.1% stabilized chlorine dioxide
- Unflavored Oral Rinse-Placebo Then Test-Unflavored Oral Rinse: CloSYS unflavored rinse containing NO 0.1% stabilized chlorine dioxide
  Unflavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Unflavored Rinse then CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide
Period: First Sequence (3 Weeks)
Arm/Group | Test-Unflavored Rinse Then Placebo-Unflavored Rinse | Test-Flavored Rinse Then Placebo-Flavored Rinse | Flavored Oral Rinse-Placebo Then Test-Flavored Rinse | Unflavored Oral Rinse-Placebo Then Test-Unflavored Oral Rinse
Started | 23 | 26 | 25 | 25
Completed | 22 | 23 | 23 | 23
Not Completed | 1 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 2
Period: Washout (2 Weeks)
Arm/Group | Test-Unflavored Rinse Then Placebo-Unflavored Rinse | Test-Flavored Rinse Then Placebo-Flavored Rinse | Flavored Oral Rinse-Placebo Then Test-Flavored Rinse | Unflavored Oral Rinse-Placebo Then Test-Unflavored Oral Rinse
Started | 22 | 23 | 23 | 23
Completed | 22 | 23 | 23 | 23
Not Completed | 0 | 0 | 0 | 0
Period: Second Sequence (3 Weeks)
Arm/Group | Test-Unflavored Rinse Then Placebo-Unflavored Rinse | Test-Flavored Rinse Then Placebo-Flavored Rinse | Flavored Oral Rinse-Placebo Then Test-Flavored Rinse | Unflavored Oral Rinse-Placebo Then Test-Unflavored Oral Rinse
Started | 22 | 23 | 23 | 23
Completed | 22 | 23 | 23 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test-Unflavored Rinse Then Placebo Unflavored Rinse: CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Unflavored Rinse: Subjects in Test group will receive ClōSYS® Unflavored Rinse then CloSYS unflavored rinse containing NO 0.1% stabilized chlorine dioxide.
- Test-Flavored Rinse Then Placebo Flavored Rinse: CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Flavored Rinse: Subjects in Test group will receive ClōSYS® Flavored Rinse then CloSYS mint flavored rinse containing NO 0.1% stabilized chlorine dioxide.
- Flavored Oral Rinse-Placebo Then Test-Flavored Rinse: CloSYS mint flavored rinse containing NO 0.1% stabilized chlorine dioxide
  Flavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Flavored Rinse then CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution.
- Unflavored Oral Rinse-Placebo Then Unflavored Oral Rinse: CloSYS unflavored rinse containing NO 0.1% stabilized chlorine dioxide
  Unflavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Unflavored Rinse then CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution.
- Total: Total of all reporting groups
Arm/Group | Test-Unflavored Rinse Then Placebo Unflavored Rinse | Test-Flavored Rinse Then Placebo Flavored Rinse | Flavored Oral Rinse-Placebo Then Test-Flavored Rinse | Unflavored Oral Rinse-Placebo Then Unflavored Oral Rinse | Total
Number analyzed (Participants) | 23 | 26 | 25 | 25 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 25 | 25 | 99
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 14 | 14 | 66
  Male | 5 | 6 | 11 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 20 | 16 | 16 | 68
  Not Hispanic or Latino | 7 | 6 | 9 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 20 | 23 | 23 | 20 | 86
  More than one race | 1 | 1 | 1 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 25 | 25 | 99

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Malodor as Measured by Organoleptic Score
Description: A 6-level organoleptic score from 0 - 5 will be used. Score of 0 indicating malodor cannot be detected and score of 5 indicating very strong malodor.
Time Frame: Weekly for three weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Test-Unflavored Rinse Then Placebo Unflavored Rinse: CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Unflavored Rinse: Subjects in Test group will receive ClōSYS® Unflavored Rinse then Placebo Unflavored rinse
- Test-Flavored Rinse Then Placebo Flavored Rinse: CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Flavored Rinse: Subjects in Test group will receive ClōSYS® Flavored Rinse then Placebo Flavored Rinse
- Flavored Oral Rinse-Placebo Then Test Flavored Oral Rinse: CloSYS mint flavored rinse containing NO 0.1% stabilized chlorine dioxide
  Flavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Flavored Rinse then Test Flavored Oral Rinse
- Unflavored Oral Rinse-Placebo Then Test Unflavored Oral Rinse: CloSYS unflavored rinse containing NO 0.1% stabilized chlorine dioxide
  Unflavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Unflavored Rinse
Arm/Group | Test-Unflavored Rinse Then Placebo Unflavored Rinse | Test-Flavored Rinse Then Placebo Flavored Rinse | Flavored Oral Rinse-Placebo Then Test Flavored Oral Rinse | Unflavored Oral Rinse-Placebo Then Test Unflavored Oral Rinse
Number analyzed (Participants) | 23 | 23 | 23 | 24
score on a scale
  Baseline 1 | 3.58 (0.67) | 3.60 (0.63) | 3.63 (0.62) | 3.65 (0.66)
  Visit 1 | 2.93 (0.40) | 2.19 (0.51) | 3.03 (0.64) | 2.29 (0.65)
  Visit 2 | 2.39 (0.61) | 1.45 (0.51) | 2.73 (0.60) | 1.81 (.58)
  Visit 3 | 2.30 (.67) | 1.15 (0.37) | 2.65 (0.56) | 1.40 (.61)
  Baseline-2 | 3.28 (0.52) | 3.25 (0.52) | 3.05 (0.38) | 3.21 (0.52)
  Visit 1-2 | 3.00 (0.35) | 2.08 (0.56) | 2.89 (0.47) | 2.08 (0.74)
  Visit 2-2 | 2.91 (0.35) | 1.48 (0.60) | 2.83 (0.50) | 1.47 (0.63)
  Visit 3-2 | 2.90 (0.35) | 1.25 (0.47) | 2.83 (0.50) | 1.34 (0.60)
Statistical Analysis 1: Comparison: Test-Flavored Rinse Then Placebo Flavored Rinse vs Flavored Oral Rinse-Placebo Then Test Flavored Oral Rinse; Test Flavored Rinse, Placebo Flavored Rinse; Test type: Superiority; p < 0.00001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Test-Unflavored Rinse Then Placebo Unflavored Rinse vs Unflavored Oral Rinse-Placebo Then Test Unflavored Oral Rinse; Test Unflavored Rinse, Placebo Unflavored Rinse; Test type: Superiority; p < 0.00001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 weeks for each intervention, 2 weeks for washout
Groups:
- Test-Unflavored Rinse: CloSYS unflavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Unflavored Rinse: Subjects in Test group will receive ClōSYS® Unflavored Rinse
- Test-Flavored Rinse: CloSYS mint-flavored rinse containing 0.1% stabilized chlorine dioxide (sodium chlorite) in an aqueous solution
  ClōSYS® Flavored Rinse: Subjects in Test group will receive ClōSYS® Flavored Rinse
- Flavored Oral Rinse-Placebo: CloSYS mint flavored rinse containing NO 0.1% stabilized chlorine dioxide
  Flavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Flavored Rinse
- Unflavored Oral Rinse-Placebo: CloSYS unflavored rinse containing NO 0.1% stabilized chlorine dioxide
  Unflavored Oral Rinse - Placebo: Subjects in Placebo group will receive Placebo Unflavored Rinse
Arm/Group | Test-Unflavored Rinse | Test-Flavored Rinse | Flavored Oral Rinse-Placebo | Unflavored Oral Rinse-Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51 | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51 | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51 | 0/51 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03160573/Prot_SAP_000.pdf